CLINICAL TRIAL: NCT05298163
Title: Effects of Calcitriol on Podocytes in Diabetic Kidney Disease Patients: Assessment of Urine Podocin, Urine Nephrin, Urine Interleukin-6, Urine KIM-1, Plasma Renin, and Albuminuria
Brief Title: The Effects of Calcitriol on Biomarkers in Diabetic Kidney Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pringgodigdo Nugroho, MD, Staff of Nephrology and Hypertension Division, Internal Medicine Department, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-176/UN2.F1/ETIK/2022
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Podocin; Nephrin; Calcitriol; Tubular injury; Podocyte injury
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Drug: Calcitriol The intervention group will be given calcitriol at a dose of 0.25 mcg/day for six months in the form of capsules that have been marked and numbered. The drugs will be taken through the RSCM pharmacy once a month during visit and the allocation will be given using drug labels that are sealed and packaged identically.
  Interventions: Drug: Calcitriol capsules
- Placebo Group (Active Comparator): Drug: Placebo oral The placebo drug will be given for six months in the form of capsules that have been marked and numbered. The drugs will be taken through the RSCM pharmacy once a month during visit and the allocation will be given using drug labels that are sealed and packaged identically.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitriol capsules — Calcitriol under the name of Oscal, 0.25 mcg/day (minimum dose) will be given for 6 months, starting at the day of the time when inclusion criteria have been met.
  Other Names: Oscal
  Arms: Intervention Group
Drug: Placebo — One placebo capsule matching the active drug will be given per day for 6 months, starting at the day of the time when inclusion criteria have been met
  Arms: Placebo Group

SUMMARY:
Diabetic Kidney Disease (DKD) is a complication that occurs due to poor glycemic control over a long period. The decrease or loss of podocytes is an important index in determining the degree of glomerular damage. Previous studies in patients with DKD reported that vitamin D administration can improve their renal function through several mechanisms. However, there is still little evidence available regarding the effects of calcitriol on biomarkers of DKD. This trial is a double-blind randomized controlled trial to assess the effect of calcitriol in DKD patients through several biomarkers which reflect pathomechanism in DKD. Those biomarkers include urinary podocin, urinary nephrin, urinary KIM-1, urinary IL-6, plasma renin, and albuminuria.

The primary outcome is any improvement on podocyte markers, tubular markers, kidney inflammation parameters, plasma renin, and albuminuria between calcitriol and placebo groups. Secondary outcomes include the relation between each marker and the side effects of intervention therapy.

DETAILED DESCRIPTION:
Diabetic Kidney Disease (DKD) is a complication that occurs due to poor glycemic control over a long period. The decrease or loss of podocytes is an important index in determining the degree of glomerular damage. Albuminuria and estimated glomerular filtration rate (eGFR) are currently used as the marker of DKD. However, these markers may not directly measure renal tissue injury. Thus, investigating novel biomarkers, particularly podocyte-associated biomarkers, is needed to predict DKD. Previous studies in patients with DKD reported that vitamin D administration can improve their renal function. of the various types of vitamin D, there is still little evidence available regarding the effects of calcitriol on biomarkers of DKD. Therefore, this study aimed to determine the effect of calcitriol on podocyte damage markers, tubular injury markers, kidney inflammation parameter, plasma renin, dan albuminuria in DKD patients.

This study is a double-blind randomized controlled clinical trial to assess the effect of calcitriol in DKD patients through several markers including albuminuria. Podocyte damage is characterized by urinary podocin and urinary nephrin, tubular marker injury is characterized by urinary KIM-1, kidney inflammation is represented by urinary IL-6, hemodynamic is represented by plasma renin.

The primary outcome is any improvement on those markers between calcitriol and placebo groups. And the secondary outcomes include the relation between each marker and the side effects of intervention therapy.

ELIGIBILITY:
Inclusion Criteria:

* Controlled type 2 diabetes mellitus with HbA1C at least <8% and albuminuria (UACR>30 mg/mmol)
* Estimated Glomerular Filtration Rate (eGFR) >45 ml/min/1.73 m2
* Agree to participate in the research

Exclusion Criteria:

* Uncontrolled hypertension with routine Angiotensin-converting-enzyme inhibitors (ACEi) or Angiotensin II receptor blockers (ARBs) treatment
* Hypercalcemia (total serum Ca level >10/5 mg/dL)
* Hyperphosphatemia (total serum phosphate level >5 mg/dL)
* Hypersensitivity to calcitriol
* Suffering from other diseases that cause proteinuria
* Acute diseases
* Smoker or previous smoking history
* Taking medications or suplements that can affect calcitriol metabolism (thiazide, digoxin, anti-convulsant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Urinary podocin | 6 months
  Marker of podocyte injury, will be measured before, during, and after treatment
Urinary nephrin | 6 months
  Marker of podocyte injury, will be measured before, during, and after treatment
Urinary KIM-1 | 6 months
  Marker of tubular injury, will be measured before, during, and after treatment
Urinary IL-6 | 6 months
  Marker of kidney inflammation, will be measured before, during, and after treatment
Plasma renin | 6 months
  Marker of hemodynamic pathway, will be measured before, during, and after treatment
Albuminuria | 6 months
  Marker of glomerular damage, will be measured before, during, and after treatment

SECONDARY OUTCOMES:
Calcium level | 6 months
  Will be measured monthly

CONTACTS AND LOCATIONS:
Overall Officials: Pringgodigdo Nugroho, MD, Principal Investigator — Division of Nephrology Hypertension, Department of Internal Medicine, Faculty of Medicine, Universitas Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin YC, Chang YH, Yang SY, Wu KD, Chu TS. Update of pathophysiology and management of diabetic kidney disease. J Formos Med Assoc. 2018 Aug;117(8):662-675. doi: 10.1016/j.jfma.2018.02.007. Epub 2018 Mar 2. PMID 29486908
- [Background] Gheith O, Farouk N, Nampoory N, Halim MA, Al-Otaibi T. Diabetic kidney disease: world wide difference of prevalence and risk factors. J Nephropharmacol. 2015 Oct 9;5(1):49-56. eCollection 2016. PMID 28197499
- [Background] Zylka A, Dumnicka P, Kusnierz-Cabala B, Gala-Bladzinska A, Ceranowicz P, Kucharz J, Zabek-Adamska A, Maziarz B, Drozdz R, Kuzniewski M. Markers of Glomerular and Tubular Damage in the Early Stage of Kidney Disease in Type 2 Diabetic Patients. Mediators Inflamm. 2018 Aug 9;2018:7659243. doi: 10.1155/2018/7659243. eCollection 2018. PMID 30158836
- [Background] Kravets I, Mallipattu SK. The Role of Podocytes and Podocyte-Associated Biomarkers in Diagnosis and Treatment of Diabetic Kidney Disease. J Endocr Soc. 2020 Mar 5;4(4):bvaa029. doi: 10.1210/jendso/bvaa029. eCollection 2020 Apr 1. PMID 32232184
- [Background] Garg P. A Review of Podocyte Biology. Am J Nephrol. 2018;47 Suppl 1:3-13. doi: 10.1159/000481633. Epub 2018 May 31. PMID 29852492
- [Background] Sekulic M, Pichler Sekulic S. A compendium of urinary biomarkers indicative of glomerular podocytopathy. Patholog Res Int. 2013;2013:782395. doi: 10.1155/2013/782395. Epub 2013 Nov 13. PMID 24327929
- [Background] Kostovska I, Tosheska-Trajkovska K, Topuzovska S, Cekovska S, Spasovski G, Kostovski O, Labudovic D. Urinary nephrin is earlier, more sensitive and specific marker of diabetic nephropathy than microalbuminuria. J Med Biochem. 2020 Jan 10;39(1):83-90. doi: 10.2478/jomb-2019-0026. PMID 32549781
- [Background] Jim B, Ghanta M, Qipo A, Fan Y, Chuang PY, Cohen HW, Abadi M, Thomas DB, He JC. Dysregulated nephrin in diabetic nephropathy of type 2 diabetes: a cross sectional study. PLoS One. 2012;7(5):e36041. doi: 10.1371/journal.pone.0036041. Epub 2012 May 17. PMID 22615747
- [Background] Martin CE, Jones N. Nephrin Signaling in the Podocyte: An Updated View of Signal Regulation at the Slit Diaphragm and Beyond. Front Endocrinol (Lausanne). 2018 Jun 5;9:302. doi: 10.3389/fendo.2018.00302. eCollection 2018. PMID 29922234
- [Background] Zhang W, Wang W, Yu H, Zhang Y, Dai Y, Ning C, Tao L, Sun H, Kellems RE, Blackburn MR, Xia Y. Interleukin 6 underlies angiotensin II-induced hypertension and chronic renal damage. Hypertension. 2012 Jan;59(1):136-44. doi: 10.1161/HYPERTENSIONAHA.111.173328. Epub 2011 Nov 7. PMID 22068875
- [Background] Marquez E, Riera M, Pascual J, Soler MJ. Renin-angiotensin system within the diabetic podocyte. Am J Physiol Renal Physiol. 2015 Jan 1;308(1):F1-10. doi: 10.1152/ajprenal.00531.2013. Epub 2014 Oct 22. PMID 25339703
- [Background] Wang Y, Deb DK, Zhang Z, Sun T, Liu W, Yoon D, Kong J, Chen Y, Chang A, Li YC. Vitamin D receptor signaling in podocytes protects against diabetic nephropathy. J Am Soc Nephrol. 2012 Dec;23(12):1977-86. doi: 10.1681/ASN.2012040383. Epub 2012 Nov 2. PMID 23123403
- [Background] Guo J, Lu C, Zhang F, Yu H, Zhou M, He M, Wang C, Zhao Z, Liu Z. VDR Activation Reduces Proteinuria and High-Glucose-Induced Injury of Kidneys and Podocytes by Regulating Wnt Signaling Pathway. Cell Physiol Biochem. 2017;43(1):39-51. doi: 10.1159/000480315. Epub 2017 Aug 24. PMID 28848172
- [Background] Yang S, Li A, Wang J, Liu J, Han Y, Zhang W, Li YC, Zhang H. Vitamin D Receptor: A Novel Therapeutic Target for Kidney Diseases. Curr Med Chem. 2018;25(27):3256-3271. doi: 10.2174/0929867325666180214122352. PMID 29446731
- [Background] Lei M, Liu Z, Guo J. The Emerging Role of Vitamin D and Vitamin D Receptor in Diabetic Nephropathy. Biomed Res Int. 2020 Jul 11;2020:4137268. doi: 10.1155/2020/4137268. eCollection 2020. PMID 32766307
- [Derived] Nugroho P, Lydia A, Soewondo P, Suhardjono, Timan IS, Harimurti K, Ali Z. Modulation of renal inflammation and tubular injury by calcitriol in patients with early diabetic kidney disease: a randomized controlled trial. Ann Med. 2025 Dec;57(1):2577271. doi: 10.1080/07853890.2025.2577271. Epub 2025 Oct 27. PMID 41145267